CLINICAL TRIAL: NCT03317080
Title: A Study of the Value of Dynamic Monitoring Circulating Tumor DNA in Patients With Lung Cancer for Post-Operative Evaluation,Therapy Response Assessment,Relapse Prediction and Defining Molecular Phenotypes.
Brief Title: Dynamic Monitoring Circulating Tumor DNA in Surgical Patients With Lung Cancer
Acronym: LUNGCA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: West China Hospital (Other)
Collaborators: GeneCast Biotechnology Co., Ltd. (Industry); Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Lunxu Liu, Professor and Chair of Department of Thoracic surgery, West China Hospital
Other Study IDs: TSCI003
Record Dates: First submitted 2017-10-12; First posted 2017-10-23 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Lung Cancer
Keywords: lung cancer; circulating tumor DNA; molecular classification; dynamic monitoring; next generation sequencing; diagnosis; postoperative relapse
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue,blood and plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with lung cancer: patients with stages I-III lung cancer eligible for surgery

SUMMARY:
This study aims to promote the rational use of liquid biopsy in the clinical detection of lung cancer. Lung cancer is a malignant tumor with high morbidity and mortality worldwide. The incidence of lung cancer in China is expected to increase in the next few years with the aging population and environmental pollution. Early diagnosis and effective intervention are necessary in the clinical treatment of lung cancer. Surgical resection could achieve a better prognosis for patients with early lung cancer. However, for advanced lung cancer, individualized treatment based on the pathological classification, molecular genetic characteristics, and body conditions of patients could effectively prolong the lifetime. The prevention, diagnosis, and intervention strategies for lung cancer depend on the oncology information of patients. The techniques and methods used for detecting lung cancer in clinic include imaging technology, pathological biopsy, screening of blood tumor markers, and liquid biopsy technology, which has been developed recently. The liquid biopsy can capture the oncology information, including tumor load, tumor gene mutation, and so on, from the blood of patients with cancer by detecting circulating tumor cells, tumor exosome, circulating tumor DNA, and circulating tumor RNA. Moreover, it has become an important direction for clinical tumor detection because of its noninvasiveness, convenient sampling, and potential for overcoming tumor heterogeneity. This study intends to include 400 patients with stage I-III lung cancer to research on lung cancer diagnosis, drug efficacy, surgical effect evaluation, recurrence monitoring, prognosis judgment, medication guidance, and molecular classification differentiation through the dynamic detection of blood ctDNA using the second-generation sequencing technology. The study also intends to analyze and establish the database with a large sample size.

DETAILED DESCRIPTION:
Lung cancer is a malignant tumor with high morbidity and mortality worldwide. The incidence and mortality of lung cancer in China have topped the list of malignant tumors since 2010.Early diagnosis and effective intervention are extremely important in the clinical treatment of lung cancer. Surgical resection could achieve better prognosis in patients with early lung cancer (stages IA and IB).For patients with advanced lung cancer (stages II, III, and IV), individualized treatment with molecular classification researches and the application of targeted drugs based on the pathological classification, molecular genetic characteristics, and body conditions of patients has been confirmed to effectively prolong the lifetime. However, the lack of effective and convenient detection approaches for capturing oncology information of patients, promoting early diagnosis and effective intervention of lung cancer, and ultimately improving the prognosis of lung cancer are limitations in achieving successful clinical treatment of lung cancer.

At present, methods used in clinical screening of lung cancer,including detection of serological markers, imaging technology, and biopsy ,have some limitations:in the absence of imaging evidence, the serological assessment could not be used as the evidence for diagnosis and treatment strategy alteration for lung cancer. The application of low-dose computed tomography scan for lung cancer screening shows a high false-positive rate, which is liable to require excessive medical treatment. Biopsy does greater harm to patients with lung cancer; sampling is difficult, and effective information may be missed because of tumor heterogeneity. With the development of molecular pathology in cancer research in recent years, liquid biopsy has become an important developmental direction for clinical tumor detection because of its noninvasiveness, convenient sampling, and potential for overcoming tumor heterogeneity.Liquid biopsies include the detection of circulating tumor cells (CTCs), tumor exosome (exosome), circulating tumor RNA (ctRNA), and circulating tumor DNA (ctDNA) in peripheral blood.

ctDNA is a part of circulating free DNA (cfDNA), which is released by tumor cell necrosis, apoptosis, micrometastasis, or the cleavage of CTCs and proliferated tumor cells.ctDNA includes genetic information of tumor cells, such as mutation, recombination, and deletion (15). ctDNA was approved by the European Medicines Agency in 2014 and the National Comprehensive Cancer Network Guidelines for NSCLC in 2017 as a supplement sample to assess genetic variation when tumor tissue samples were difficult to obtain. Clinical studies have shown that ctDNA can effectively reflect tumor load, malignant degree, metastasis ability, and real-time information of genetic mutation, which has a certain correlation with the genetic information of tumor tissues. Moreover, the content of cfDNA in patients with cancer was significantly higher than that in healthy people. Also, ctDNA has been used for detecting tumor load, monitoring tumor recurrence, and assessing minimal residual disease in a number of cancer types. Some studies have suggested that ctDNA can be used to estimate tumor recurrence, even before imaging. Therefore, ctDNA detection has an important value in the clinical application of lung cancer diagnosis, drug efficacy, surgical effect evaluation, recurrence monitoring, prognosis judgment, medication guidance, and molecular classification differentiation.

This study intends to include 400 patients with stage I-III lung cancer. The capture sequencing of lung cancer-related genes in peripheral blood ctDNA and tumor tissue DNA will be performed during the diagnosis and treatment process using the liquid-phase hybridization approach. Thus, the study will establish a large sample size database of the genetic variants in patients with lung cancer during the diagnosis and treatment process, and promoted the development of an individualized diagnostic model of the lung cancer population. The patients with lung cancer undergoing surgery will be followed up, and the plasma concentration of cfDNA and genetic mutation of ctDNA will be detected to evaluate the postoperative residual cancer, monitor tumor recurrence, and timely guide the clinical treatment and intervention. The molecular classification differentiation analysis and screening of tumor recurrence-related genetic mutations will be performed after the surgery and during the course of disease progression to provide the referential clinical research model and ideas for the application of ctDNA detection-based liquid biopsy technique in tumor therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage I-III lung cancer who are eligible for surgery(with no restriction of age, gender, or smoking history).
2. ECOG score:0-1.
3. Patients in the group will be allowed to collect whole blood or tissue samples at specific time points.
4. Patients will be regularly tested according to the doctor's advice.
5. Signed informed consent.

Exclusion Criteria:

1. The tumor manifests as pure GGO on chest CT scan.
2. Patients for surgical biopsy.
3. Patients with serious mental disease.
4. Surgery is contraindicated for any reason.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with stage I-III lung cancer eligible for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-09-27 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
recurrence-free survival | up to 36 months
  from the date of surgery until the date of first verified recurrence or death from any cause

SECONDARY OUTCOMES:
overall survival | up to 36 months
  from the date of surgery until the date of death from any cause
heterogeneity of lung cancer | up to 36 months
  the relationship between heterogeneity of lung cancer and clinical results following surgery and adjuvant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Lunxu Liu, M.D.,Ph.D., Principal Investigator — Department of Thoracic Surgery, West China Hospital, Sichuan University
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ren JS, Masuyer E, Ferlay J. Global estimates of cancer prevalence for 27 sites in the adult population in 2008. Int J Cancer. 2013 Mar 1;132(5):1133-45. doi: 10.1002/ijc.27711. Epub 2012 Jul 26. PMID 22752881
- [Background] Tsoi KK, Hirai HW, Chan FC, Griffiths S, Sung JJ. Cancer burden with ageing population in urban regions in China: projection on cancer registry data from World Health Organization. Br Med Bull. 2017 Jan 1;121(1):83-94. doi: 10.1093/bmb/ldw050. PMID 27913398
- [Background] Guo Y, Zeng H, Zheng R, Li S, Pereira G, Liu Q, Chen W, Huxley R. The burden of lung cancer mortality attributable to fine particles in China. Sci Total Environ. 2017 Feb 1;579:1460-1466. doi: 10.1016/j.scitotenv.2016.11.147. Epub 2016 Nov 29. PMID 27913022
- [Background] Chansky K, Sculier JP, Crowley JJ, Giroux D, Van Meerbeeck J, Goldstraw P; International Staging Committee and Participating Institutions. The International Association for the Study of Lung Cancer Staging Project: prognostic factors and pathologic TNM stage in surgically managed non-small cell lung cancer. J Thorac Oncol. 2009 Jul;4(7):792-801. doi: 10.1097/JTO.0b013e3181a7716e. PMID 19458556
- [Background] Perez-Ramirez C, Canadas-Garre M, Robles AI, Molina MA, Faus-Dader MJ, Calleja-Hernandez MA. Liquid biopsy in early stage lung cancer. Transl Lung Cancer Res. 2016 Oct;5(5):517-524. doi: 10.21037/tlcr.2016.10.15. PMID 27826533
- [Background] Groome PA, Bolejack V, Crowley JJ, Kennedy C, Krasnik M, Sobin LH, Goldstraw P; IASLC International Staging Committee; Cancer Research and Biostatistics; Observers to the Committee; Participating Institutions. The IASLC Lung Cancer Staging Project: validation of the proposals for revision of the T, N, and M descriptors and consequent stage groupings in the forthcoming (seventh) edition of the TNM classification of malignant tumours. J Thorac Oncol. 2007 Aug;2(8):694-705. doi: 10.1097/JTO.0b013e31812d05d5. PMID 17762335
- [Background] Su C, Meyer M, Pirker R, Voigt W, Shi J, Pilz L, Huber RM, Wu Y, Wang J, He Y, Wang X, Zhang J, Zhi X, Shi M, Zhu B, Schoenberg SS, Henzler T, Manegold C, Zhou C, Roessner ED. From diagnosis to therapy in lung cancer: management of CT detected pulmonary nodules, a summary of the 2015 Chinese-German Lung Cancer Expert Panel. Transl Lung Cancer Res. 2016 Aug;5(4):377-88. doi: 10.21037/tlcr.2016.07.09. PMID 27652202
- [Background] Rolfo C, Castiglia M, Hong D, Alessandro R, Mertens I, Baggerman G, Zwaenepoel K, Gil-Bazo I, Passiglia F, Carreca AP, Taverna S, Vento R, Santini D, Peeters M, Russo A, Pauwels P. Liquid biopsies in lung cancer: the new ambrosia of researchers. Biochim Biophys Acta. 2014 Dec;1846(2):539-46. doi: 10.1016/j.bbcan.2014.10.001. Epub 2014 Oct 16. PMID 25444714
- [Background] Stroun M, Lyautey J, Lederrey C, Olson-Sand A, Anker P. About the possible origin and mechanism of circulating DNA apoptosis and active DNA release. Clin Chim Acta. 2001 Nov;313(1-2):139-42. doi: 10.1016/s0009-8981(01)00665-9. PMID 11694251
- [Background] van der Vaart M, Pretorius PJ. The origin of circulating free DNA. Clin Chem. 2007 Dec;53(12):2215. doi: 10.1373/clinchem.2007.092734. No abstract available. PMID 18267930
- [Background] van der Vaart M, Pretorius PJ. Circulating DNA. Its origin and fluctuation. Ann N Y Acad Sci. 2008 Aug;1137:18-26. doi: 10.1196/annals.1448.022. PMID 18837919
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Schwarzenbach H, Hoon DS, Pantel K. Cell-free nucleic acids as biomarkers in cancer patients. Nat Rev Cancer. 2011 Jun;11(6):426-37. doi: 10.1038/nrc3066. Epub 2011 May 12. PMID 21562580
- [Background] Leon SA, Shapiro B, Sklaroff DM, Yaros MJ. Free DNA in the serum of cancer patients and the effect of therapy. Cancer Res. 1977 Mar;37(3):646-50. PMID 837366
- [Background] Ueda M, Iguchi T, Masuda T, Nakahara Y, Hirata H, Uchi R, Niida A, Momose K, Sakimura S, Chiba K, Eguchi H, Ito S, Sugimachi K, Yamasaki M, Suzuki Y, Miyano S, Doki Y, Mori M, Mimori K. Somatic mutations in plasma cell-free DNA are diagnostic markers for esophageal squamous cell carcinoma recurrence. Oncotarget. 2016 Sep 20;7(38):62280-62291. doi: 10.18632/oncotarget.11409. PMID 27556701
- [Background] Tie J, Wang Y, Tomasetti C, Li L, Springer S, Kinde I, Silliman N, Tacey M, Wong HL, Christie M, Kosmider S, Skinner I, Wong R, Steel M, Tran B, Desai J, Jones I, Haydon A, Hayes T, Price TJ, Strausberg RL, Diaz LA Jr, Papadopoulos N, Kinzler KW, Vogelstein B, Gibbs P. Circulating tumor DNA analysis detects minimal residual disease and predicts recurrence in patients with stage II colon cancer. Sci Transl Med. 2016 Jul 6;8(346):346ra92. doi: 10.1126/scitranslmed.aaf6219. PMID 27384348